CLINICAL TRIAL: NCT01081795
Title: A Placebo-Controlled Dose-Finding Study of JNS019 (Topiramate) in Migraine Patients
Brief Title: A Dose-Finding Study of Topiramate (JNS019) in Participants With Migraine
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR013681; JNS019-JPN-02
Record Dates: First submitted 2010-03-04; First posted 2010-03-05 (Estimated); Results first posted 2013-05-06 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-06

CONDITIONS: Migraine
Keywords: Topiramate; Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Topiramate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Topiramate (JNS019) 50 mg (Experimental): In titration period, topiramate 25 milligram (mg) tablet will be given once daily in evening orally for 7 days; then topiramate 25 mg tablet twice daily orally from Day 8 to Day 14; then topiramate 25 mg tablet twice daily along with matching placebo tablet once daily in the evening orally from Day 15 to Day 21; then topiramate 25 mg tablet along with matching placebo tablet twice daily orally from Day 22 to Day 28 and will be continued further for 18 weeks in the fixed dose period.
  Interventions: Drug: Topiramate; Drug: Placebo
- Topiramate 100 mg (Experimental): In titration period, topiramate 25 mg tablet will be given once daily in the evening orally for 7 days; then topiramate 25 mg tablet twice daily orally from Day 8 to Day 14; then topiramate 25 mg tablet twice daily (1 tablet in the morning and 2 tablets in the evening) orally from Day 15 to Day 21; then 2 topiramate 25 mg tablets twice daily orally from Day 22 to Day 28 and will be continued further for 18 weeks in the fixed dose period.
  Interventions: Drug: Topiramate
- Placebo (Placebo Comparator): In titration period, matching placebo tablet will be given once daily in evening orally for 7 days; followed by matching placebo tablet twice daily orally from Day 8 to Day 14; followed by matching placebo tablet twice daily (1 tablet in the morning and 2 tablets in the evening) orally from Day 15 to Day 21; followed by 2 matching placebo tablets twice orally from Day 22 to Day 28 and will becontinued further for 18 weeks in the fixed dose period.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Topiramate — In the titration period, topiramate 25-mg tablet once daily orally for 1 week, the dose will be increased by 1 tablet every week up to twice daily for a total of 4 weeks so that the total daily dose given is 50 mg or 100mg. The dose given in the final titration week will be continued for further 18 weeks (fixed dose period).
  Arms: Topiramate (JNS019) 50 mg; Topiramate 100 mg
Drug: Placebo — In the titration period, matching placebo tablet once daily orally for 1 week, the dose will be increased by 1 tablet every week up to twice daily for a total of 4 weeks. The dose given in the final titration week will be continued for further 18 weeks (fixed dose period).
  Arms: Placebo; Topiramate (JNS019) 50 mg

SUMMARY:
The purpose of this study is to determine a recommended dose of topiramate in participants with migraine (type of severe headache that occurs periodically and is often associated with nausea, vomiting, and constipation or diarrhea), to verify the superiority (statistically more effective) of the drug to placebo (an inactive substance that is compared with a drug to test whether the drug has a real effect in a clinical trial), and to assess if a same therapeutic effect can be observed between this study and overseas Caucasian clinical studies.

DETAILED DESCRIPTION:
This study is a multicenter (more than 1 site), placebo-controlled (compared to placebo), randomized (participants assigned study drug by chance), double-blind (neither the participant nor the physician know the assigned study drug), parallel-group comparison (comparison for each group at the same time) study. The study period consists of 4 phases: the observation phase, double-blind phase, exit period and follow-up period. After the double-blind phase, the participants will be transferred to the continuous treatment study. The observation phase which is started after informed consent consists of the washout period (non-treatment period with migraine preventive medication: at least 2 weeks) and baseline determination period (at least 4 weeks). The participants who complete the observation phase and meet the inclusion criteria will be randomly assigned to the topiramate 50 milligram (mg) group, topiramate 100-mg group or placebo group after registration. The double-blind phase consists of the titration period (dose-escalation, 4 weeks) and fixed-dose period (18 weeks). In the titration period, starting from 1 topiramate 25-mg tablet or 1 topiramate 25-mg placebo tablet once daily (1 tablet in the evening), the dose will be increased by 1 tablet every week up to twice daily (2 tablets in the morning, 2 tablets in the evening). After that, the twice-daily treatment (2 tablets in the morning, 2 tablets in the evening) will be continued for 7 days from Day 22 to Day 28. In the fixed-dose period, the topiramate 25-mg tablets or topiramate 25-mg placebo tablets at the same dose as that in the final treatment in titration period will be continued. The participants who are not transferred to the continuous treatment study after completion of the double-blind phase or after discontinuation during the double-blind phase will be transferred to the exit period (up to 1 week).The participants who complete the exit period will be transferred to the follow-up period, and a follow-up of the participant's safety and headache symptoms such as the migraine period rate will be conducted for 4 weeks after the completion of investigational treatment. Meanwhile, the participants who complete the double-blind phase or those who discontinue the study at Week 4 or later in the fixed-dose period during the double-blind phase due to lack of efficacy and give consent to transfer to the continuous treatment study will be transferred to the transfer period (up to 3 weeks) under blind conditions.

ELIGIBILITY:
Inclusion Criteria:

* Participants who meet the Second Edition of the International Classification of Headache Disorders (ICHD-II), 1.1 Migraine without aura or 1.2 Migraine with aura over at least 6 months before the time of informed consent
* Participants who had an average of no more than 8 migraine attacks per month during 3 months before informed consent and an average of no more than 14 headache (migraine and non-migraine) days
* Participants whose number of migraine attacks during the baseline determination period (28 days) is 3 to 12 according to the 24-hour rule and number of headache days (migraine and non-migraine) is no more than 14
* Participants who took no migraine preventive medications over 2 weeks before informed consent, or who can take at least 2-week washout period before baseline determination period if they are taking migraine preventive medications
* Female participants must be postmenopausal, surgically sterile, abstinent, or can take adequate contraceptive measures after informed consent and continue it to the completion of investigational treatment

Exclusion Criteria:

* Participants who cannot distinguish between migraine and non-migraine headache
* Participants with headache other than those described in the ICHD-II, 1.1 Migraine without aura, 1.2 Migraine with aura, 2. Tension headache or 11.5 Sinus headache
* If the participant has received drug therapies for prevention of migraine, the discontinued preventive therapies due to insufficient efficacy should be at least three types
* Participants who excessively took medications for migraine attacks such as analgesics (drug used to control pain) as medications to be taken as needed within 3 months before informed consent
* Participants who have taken topiramate (test drug in this study) in the past

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 387 (Actual)
Dates: Start 2007-04; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K. Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (29):
- Japan (29):
  - Bunkyō City
  - Chitose
  - Hachiōji
  - Iruma
  - Isehara
  - Kagoshima
  - Kamogawa
  - Kitakyushu
  - Kobe
  - Kumamoto
  - Kyoto
  - Minato
  - Morioka
  - Nagoya
  - Nishinomiya
  - Numakunai
  - Sagamihara
  - Sapporo
  - Shimotsuga
  - Shinjuku
  - Shinjuku-Ku
  - Shizuoka
  - Suginami-Ku
  - Tokyo
  - Toyama
  - Toyonaka
  - Ube
  - Yokohama
  - Yonago

RESULTS

PARTICIPANT FLOW:
Groups:
- Topiramate (JNS019) 50 mg: In titration period, topiramate 25 milligram (mg) tablet once daily in evening orally for 7 days; then topiramate 25 mg tablet twice daily orally from Day 8 to Day 14; then topiramate 25 mg tablet twice daily along with matching placebo tablet once daily in the evening orally from Day 15 to Day 21; then topiramate 25 mg tablet along with matching placebo tablet twice daily orally from Day 22 to Day 28 and continued further for 18 weeks in the fixed dose period
- Topiramate 100 mg: In titration period, topiramate 25 mg tablet once daily in the evening orally for 7 days; then topiramate 25 mg tablet twice daily orally from Day 8 to Day 14; then topiramate 25 mg tablet twice daily (1 tablet in the morning and 2 tablets in the evening) orally from Day 15 to Day 21; then 2 topiramate 25 mg tablets twice daily orally from Day 22 to Day 28 and continued further for 18 weeks in the fixed dose period
- Placebo: In titration period, matching placebo tablet once daily in evening orally for 7 days; followed by matching placebo tablet twice daily orally from Day 8 to Day 14; followed by matching placebo tablet twice daily (1 tablet in the morning and 2 tablets in the evening) orally from Day 15 to Day 21; followed by 2 matching placebo tablets twice daily orally from Day 22 to Day 28 and continued further for 18 weeks in the fixed dose period
Period: Overall Study
Arm/Group | Topiramate (JNS019) 50 mg | Topiramate 100 mg | Placebo
Started | 130 | 130 | 127
Completed | 97 | 95 | 97
Not Completed | 33 | 35 | 30
Not completed — Adverse Event | 18 | 23 | 6
Not completed — Lack of Efficacy | 7 | 5 | 19
Not completed — Subject's schedule | 1 | 1 | 2
Not completed — Revocation of informed consent | 2 | 0 | 0
Not completed — Ineligible for participation | 1 | 0 | 0
Not completed — Use of a prohibited concomitant drug | 1 | 1 | 1
Not completed — Using drug with restricted days of use | 2 | 3 | 2
Not completed — Other | 1 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Topiramate (JNS019) 50 mg | Topiramate 100 mg | Placebo | Total
Number analyzed (Participants) | 130 | 130 | 127 | 387
Age Continuous [Mean (Standard Deviation); unit: Years] | 40.4 (9.30) | 39.5 (9.25) | 41.2 (9.10) | 40.3 (9.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 100 | 103 | 306
  Male | 27 | 30 | 24 | 81

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Monthly Migraine Attacks (According to 24-Hour Rule) Through Month 6
Description: As per 24-hour rule, if symptom of pain due to migraine continues for more than 24 hours, it should be considered as 2 or more migraine attacks considering the maximum duration up to 24 hours. If the interval between latest migraine attack (ending time) and previous migraine attack (onset time) is less than 24 hours, 2 migraine attacks should be considered as 1 migraine attack. If the onset of migraine was prevented by a rescue drug, it should be considered as 1 migraine attack even if aura had started. Mean change was calculated by subtracting baseline value from the mean of 6 months value.
Time Frame: Baseline (28 days before randomization) through Month 6
Population: Full analysis set (FAS) included all participants randomly assigned to study treatment excluding those who did not meet eligibility criteria, did not receive study treatment at all and did not provide any efficacy data after randomization.
Measure: Mean (Standard Deviation); unit: Migraine attacks
Arm/Group | Topiramate (JNS019) 50 mg | Topiramate 100 mg | Placebo
Number analyzed (Participants) | 130 | 130 | 127
Migraine attacks
  Baseline | 5.9 (1.79) | 6.2 (2.11) | 6.6 (2.29)
  Change at Month 6 | -0.9 (2.50) | -1.2 (2.72) | -1.0 (2.42)
Statistical Analysis 1: Comparison: Topiramate 100 mg vs Placebo; Test type: Superiority or Other; p = 0.1646, ANCOVA — Analysis of covariance (ANCOVA) method using the treatment group as the factor and using the value obtained during the baseline measurement period as the covariate was used; Least Square (LS) mean difference = -0.4, 95% CI 2-sided [-1.0 to 0.2]
Statistical Analysis 2: Comparison: Topiramate (JNS019) 50 mg vs Placebo; Test type: Superiority or Other; p = 0.4479, ANCOVA — ANCOVA method using the treatment group as the factor and using the value obtained during the baseline measurement period as the covariate was used; LS mean difference = -0.2, 95% CI 2-sided [-0.8 to 0.4]

2. Secondary Outcome: Change From Baseline in Average Number of Monthly Migraine Attack Days at Month 1, 2, 3, 4, 5 and 6
Description: Migraine is a headache disorder with 2 subtypes: migraine without aura (at least 5 attacks lasting 4-72 hours with at least 2 following characteristics: unilateral location, pulsating quality, moderate/severe pain and either nausea/vomiting or photophobia and phonophobia) and migraine with aura (reversible focal neurological symptoms that develop over 5-20 minutes and last for less than 60 minutes); average at given month was calculated by dividing total number of migraine attack days until that month by the total number of days of assessment, multiplied by 28 (a month was equal to 28 days).
Time Frame: Baseline (28 days before randomization), Month 1, 2, 3, 4, 5 and 6
Population: The FAS included all participants randomly assigned to study treatment excluding those who did not meet eligibility criteria, did not receive study treatment at all and did not provide any efficacy data after randomization.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Topiramate (JNS019) 50 mg | Topiramate 100 mg | Placebo
Number analyzed (Participants) | 130 | 130 | 127
Days
  Baseline | 6.6 (2.21) | 7.0 (2.35) | 7.3 (2.58)
  Change at Month 1 | -0.5 (2.93) | -0.8 (3.75) | -0.4 (3.18)
  Change at Month 2 | -0.7 (2.82) | -1.1 (3.36) | -0.7 (2.83)
  Change at Month 3 | -0.9 (2.74) | -1.2 (3.27) | -0.9 (2.73)
  Change at Month 4 | -0.9 (2.73) | -1.3 (3.20) | -1.0 (2.66)
  Change at Month 5 | -1.0 (2.76) | -1.3 (3.22) | -1.0 (2.70)
  Change at Month 6 | -1.0 (2.83) | -1.3 (3.24) | -1.0 (2.72)
Statistical Analysis 1: Comparison: Topiramate 100 mg vs Placebo; Test type: Superiority or Other; p = 0.1547, ANCOVA — Month 6: ANCOVA method using the treatment group as the factor and using the value obtained during the baseline measurement period as the covariate was used; LS mean difference = -0.5, 95% CI 2-sided [-1.1 to 0.2]
Statistical Analysis 2: Comparison: Topiramate (JNS019) 50 mg vs Placebo; Test type: Superiority or Other; p = 0.2624, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS mean difference = -0.4, 95% CI 2-sided [-1.0 to 0.3]

3. Secondary Outcome: Change From Baseline in Average Number of Monthly Headache Days at Month 1, 2, 3, 4, 5 and 6
Description: Headache days were the days when at least 30-minute migraine and non-migraine headache occurred and were calculated from the headache diaries kept by the participants. Average at given month was calculated by dividing total number of headache days until that month by the total number of days of assessment, multiplied by 28 (a month was equal to 28 days).
Time Frame: Baseline (28 days before randomization), Month 1, 2, 3, 4, 5 and 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Topiramate (JNS019) 50 mg | Topiramate 100 mg | Placebo
Number analyzed (Participants) | 130 | 130 | 127
Days
  Baseline | 6.9 (2.39) | 7.4 (2.48) | 7.7 (2.77)
  Change at Month 1 | -0.6 (3.00) | -0.8 (3.69) | -0.4 (3.23)
  Change at Month 2 | -0.8 (2.88) | -1.2 (3.33) | -0.8 (2.85)
  Change at Month 3 | -1.0 (2.81) | -1.3 (3.25) | -0.9 (2.72)
  Change at Month 4 | -1.1 (2.81) | -1.4 (3.15) | -1.1 (2.64)
  Change at Month 5 | -1.1 (2.83) | -1.4 (3.17) | -1.2 (2.68)
  Change at Month 6 | -1.1 (2.89) | -1.4 (3.18) | -1.2 (2.70)
Statistical Analysis 1: Comparison: Topiramate 100 mg vs Placebo; Test type: Superiority or Other; p = 0.2464, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS mean difference = -0.4, 95% CI 2-sided [-1.0 to 0.3]
Statistical Analysis 2: Comparison: Topiramate (JNS019) 50 mg vs Placebo; Test type: Superiority or Other; p = 0.3148, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS mean difference = -0.3, 95% CI 2-sided [-1.0 to 0.3]

4. Secondary Outcome: Change From Baseline in Average Number of Monthly Migraine Attacks (According to the Diagnostic Criteria of the International Headache Society) at Month 1, 2, 3, 4, 5 and 6
Description: Migraine is a headache disorder with 2 subtypes: migraine without aura (at least 5 attacks lasting 4-72 hours with at least 2 following characteristics: unilateral location, pulsating quality, moderate/severe pain and either nausea/vomiting or photophobia and phonophobia) and migraine with aura (reversible focal neurological symptoms that develop over 5-20 minutes and last for less than 60 minutes); average at given month was calculated by dividing total number of migraine attacks until that month by the total number of days of assessment, multiplied by 28 (a month was equal to 28 days).
Time Frame: Baseline (28 days before randomization), Month 1, 2, 3, 4, 5 and 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Migraine attacks
Arm/Group | Topiramate (JNS019) 50 mg | Topiramate 100 mg | Placebo
Number analyzed (Participants) | 130 | 130 | 127
Migraine attacks
  Baseline | 4.1 (2.25) | 4.3 (2.94) | 4.2 (2.93)
  Change at Month 1 | -0.8 (2.60) | -0.4 (2.92) | -0.5 (2.37)
  Change at Month 2 | -0.9 (2.61) | -0.7 (2.75) | -0.7 (2.27)
  Change at Month 3 | -0.9 (2.56) | -0.8 (2.71) | -0.7 (2.13)
  Change at Month 4 | -1.0 (2.54) | -0.9 (2.68) | -0.8 (2.15)
  Change at Month 5 | -1.1 (2.56) | -0.9 (2.69) | -0.8 (2.18)
  Change at Month 6 | -1.1 (2.59) | -0.9 (2.68) | -0.8 (2.17)
Statistical Analysis 1: Comparison: Topiramate 100 mg vs Placebo; Test type: Superiority or Other; p = 0.8762, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS mean difference = 0.0, 95% CI 2-sided [-0.6 to 0.5]
Statistical Analysis 2: Comparison: Topiramate (JNS019) 50 mg vs Placebo; Test type: Superiority or Other; p = 0.3031, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS mean difference = -0.3, 95% CI 2-sided [-0.8 to 0.3]

5. Secondary Outcome: Change From Baseline in Monthly Migraine Attacks (According to 48-Hour Rule) at Month 1, 2, 3, 4, 5 and 6
Description: As per 48-hour rule, if the symptom of pain due to migraine continues for more than 48 hours, it should be considered as 2 or more migraine attacks considering the maximum duration up to 48 hours. If the interval between the latest migraine attack (ending time) and the previous migraine attack (onset time) is less than 48 hours, the 2 migraine attacks should be considered as 1 migraine attack. If the onset of the migraine was prevented by a rescue drug, it should be considered as 1 migraine attack even if the aura had started.
Time Frame: Baseline (28 days before randomization), Month 1, 2, 3, 4, 5 and 6
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Migraine attacks
Arm/Group | Topiramate (JNS019) 50 mg | Topiramate 100 mg | Placebo
Number analyzed (Participants) | 130 | 130 | 127
Migraine attacks
  Baseline | 4.6 (1.28) | 4.9 (1.52) | 5.1 (1.56)
  Change at Month 1 | -0.2 (1.94) | -0.6 (2.28) | -0.3 (1.93)
  Change at Month 2 | -0.5 (1.77) | -0.8 (2.03) | -0.6 (1.76)
  Change at Month 3 | -0.6 (1.73) | -0.9 (1.95) | -0.7 (1.70)
  Change at Month 4 | -0.6 (1.71) | -1.0 (1.90) | -0.7 (1.70)
  Change at Month 5 | -0.7 (1.72) | -1.0 (1.91) | -0.8 (1.71)
  Change at Month 6 | -0.7 (1.75) | -1.0 (1.92) | -0.8 (1.72)
Statistical Analysis 1: Comparison: Topiramate 100 mg vs Placebo; Test type: Superiority or Other; p = 0.1145, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS mean difference = -0.3, 95% CI 2-sided [-0.7 to 0.1]
Statistical Analysis 2: Comparison: Topiramate (JNS019) 50 mg vs Placebo; Test type: Superiority or Other; p = 0.3971, ANCOVA — [p-value comment as in outcome 2, analysis 1]; LS mean difference = -0.2, 95% CI 2-sided [-0.6 to 0.2]

6. Secondary Outcome: Change From Baseline in Migraine Attacks (According to 24-Hour Rule) Over Week 19 to Week 22 Period
Description: The change from baseline in average number of migraine attacks (as per 24-hour rule) over Week 19 to Week 22 period was calculated by subtracting the baseline value from the average value of the Week 19 to Week 22 period.
Time Frame: Baseline (28 days before randomization), Week 19 to Week 22 Period
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Migraine attacks
Arm/Group | Topiramate (JNS019) 50 mg | Topiramate 100 mg | Placebo
Number analyzed (Participants) | 130 | 130 | 127
Migraine attacks | -1.3 (0.28) | -1.2 (0.28) | -0.7 (0.28)
Statistical Analysis 1: Comparison: Topiramate 100 mg vs Placebo; Test type: Superiority or Other; p = 0.1866, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS mean difference = -0.5, 95% CI 2-sided [-1.3 to 0.3]
Statistical Analysis 2: Comparison: Topiramate (JNS019) 50 mg vs Placebo; Test type: Superiority or Other; p = 0.1507, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS mean difference = -0.6, 95% CI 2-sided [-1.4 to 0.2]

7. Secondary Outcome: Average Number of Rescue Drug Treatment Days
Description: Rescue medications are administered to participants when efficacy of study drug is not satisfactory, or effect of study drug is too great and is likely to cause a hazard to participant, or to manage an emergency situation. If an aura of migraine, a migraine attack or a non-migraine headache attack occurred during the study period, use of following rescue drugs was permitted: analgesics, non-steroidal anti-inflammatory drugs (NSAIDs), ergotamines, triptans and anti-emetics (drug used to stop vomiting). Average at baseline was calculated by dividing total number of rescue drug treatment days until baseline by the total number of days of assessment, multiplied by 28 (a month was equal to 28 days).
Time Frame: Baseline (28 days before randomization)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Topiramate (JNS019) 50 mg | Topiramate 100 mg | Placebo
Number analyzed (Participants) | 130 | 130 | 127
Days | 5.5 (2.21) | 5.7 (2.50) | 6.1 (2.43)

8. Secondary Outcome: Change From Baseline in the Average Number of Rescue Drug Treatment Days at Month 6
Description: Rescue medications are medicines that may be administered to the participants when efficacy of study drug is not satisfactory, or the effect of study drug is too great and is likely to cause a hazard to the participant, or to manage an emergency situation. If an aura of migraine, a migraine attack or a non-migraine headache attack occurred during the study period, use of following rescue drugs was permitted: analgesics, NSAIDs, ergotamines, triptans and anti-emetics. Average at Month 6 was calculated by dividing total number of rescue drug treatment days until that month by the total number of days of assessment, multiplied by 28 (a month was equal to 28 days).
Time Frame: Month 6
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Days
Arm/Group | Topiramate (JNS019) 50 mg | Topiramate 100 mg | Placebo
Number analyzed (Participants) | 130 | 130 | 127
Days | -0.8 (0.21) | -0.8 (0.21) | -0.4 (0.22)
Statistical Analysis 1: Comparison: Topiramate 100 mg vs Placebo; Test type: Superiority or Other; p = 0.1743, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS mean difference = -0.4, 95% CI 2-sided [-1.0 to 0.2]
Statistical Analysis 2: Comparison: Topiramate (JNS019) 50 mg vs Placebo; Test type: Superiority or Other; p = 0.2165, ANCOVA — [p-value comment as in outcome 1, analysis 2]; LS mean difference = -0.4, 95% CI 2-sided [-1.0 to 0.2]

9. Secondary Outcome: Percentage of Participants With Response to Study Treatment
Description: Responders were the participants who had at least 50 percent reduction in the average number of monthly migraine attacks.
Time Frame: Month 1, 2, 3, 4, 5 and 6
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Topiramate (JNS019) 50 mg | Topiramate 100 mg | Placebo
Number analyzed (Participants) | 130 | 130 | 127
Percentage of participants
  Month 1 | 10.8 | 23.1 | 11.8
  Month 2 | 16.9 | 23.1 | 14.2
  Month 3 | 14.6 | 20.8 | 9.4
  Month 4 | 15.4 | 18.5 | 14.2
  Month 5 | 15.4 | 19.2 | 14.2
  Month 6 | 15.4 | 18.5 | 13.4
Statistical Analysis 1: Comparison: Topiramate 100 mg vs Placebo; Test type: Superiority or Other; p = 0.3083, Fisher Exact — Month 6; Percentage difference = 5.1, 95% CI 2-sided [-3.8 to 14.0]
Statistical Analysis 2: Comparison: Topiramate (JNS019) 50 mg vs Placebo; Test type: Superiority or Other; p = 0.7235, Fisher Exact — Month 6; Percentage difference = 2.0, 95% CI 2-sided [-6.6 to 10.6]

10. Secondary Outcome: Short Form-36 Health Survey (SF-36) Score
Description: The SF-36 is a survey of participant health. It consists of 8 scaled scores, which are weighted sums of the questions in their section. The 8 sections are: vitality, physical functioning, bodily pain, general health perceptions, physical role functioning, emotional role functioning, social role functioning and mental health. Each item is scored on a 0-100 range so that total score ranges from 0-100 with high score indicating more favorable health state. Final evaluation was done at Day 155 or at discontinuation for those participants who discontinued before Day 155.
Time Frame: Baseline (28 days before randomization), Day 29, 85 and final evaluation (FE) (Day 155/early withdrawal [EW])
Population: The FAS included all participants randomly assigned to study treatment excluding those who did not meet eligibility criteria, did not receive study treatment at all and did not provide any efficacy data after randomization. Here 'n' signifies those participants who were evaluable for this measure at given time points.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Topiramate (JNS019) 50 mg | Topiramate 100 mg | Placebo
Number analyzed (Participants) | 130 | 130 | 127
Units on a scale
  Physical functioning: Baseline (n=130,130,127) | 53.59 (5.029) | 53.84 (8.267) | 54.17 (5.669)
  Physical functioning: Day 29 (n=127,122,125) | 53.03 (6.459) | 53.15 (7.732) | 54.26 (5.520)
  Physical functioning: Day 85 (n=111,109,121) | 53.86 (5.989) | 53.85 (7.160) | 54.47 (5.437)
  Physical functioning:FE (Day155/EW)(n=130,130,127) | 54.02 (5.606) | 53.79 (7.643) | 54.40 (5.788)
  Role-Physical: Baseline (n=130,130,127) | 46.10 (9.529) | 45.29 (11.095) | 45.86 (9.247)
  Role-Physical: Day 29 (n=127,122,125) | 44.49 (10.892) | 46.05 (11.094) | 46.35 (9.700)
  Role-Physical: Day 85 (n=111,109,121) | 45.88 (9.687) | 46.34 (10.320) | 46.95 (9.624)
  Role-Physical: FE (Day 155/EW) (n=130,130,127) | 45.21 (10.675) | 45.69 (10.384) | 46.29 (9.230)
  Bodily pain: Baseline (n=130,130,127) | 40.75 (8.822) | 41.76 (10.171) | 39.67 (9.164)
  Bodily pain: Day 29 (n=127,122,125) | 42.98 (10.029) | 44.43 (10.352) | 41.17 (9.716)
  Bodily pain: Day 85 (n=111,109,121) | 43.09 (9.450) | 44.43 (9.923) | 42.03 (8.557)
  Bodily pain: FE (Day 155/EW) (n=130,130,127) | 42.64 (8.504) | 43.82 (9.906) | 42.87 (8.776)
  General health: Baseline (n=130,130,127) | 47.56 (8.444) | 48.92 (8.571) | 47.61 (7.894)
  General health: Day 29 (n=127,122,125) | 47.30 (8.996) | 49.21 (9.176) | 49.12 (7.904)
  General health: Day 85 (n=111,109,121) | 47.48 (8.827) | 48.70 (9.857) | 49.31 (8.053)
  General health: FE (Day 155/EW) (n=130,130,127) | 47.48 (8.459) | 48.12 (9.425) | 49.86 (8.713)
  Vitality: Baseline (n=130,130,127) | 48.91 (7.754) | 49.10 (7.765) | 49.17 (8.393)
  Vitality: Day 29 (n=127,122,125) | 47.72 (8.888) | 47.59 (9.900) | 50.78 (8.579)
  Vitality: Day 85 (n=111,109,121) | 48.45 (9.484) | 48.04 (9.375) | 49.40 (8.790)
  Vitality: FE (Day 155/EW) (n=130,130,127) | 47.73 (9.625) | 47.66 (9.850) | 50.34 (8.683)
  Social functioning: Baseline (n=130,130,127) | 47.62 (9.342) | 47.98 (10.108) | 47.82 (10.095)
  Social functioning: Day 29 (n=127,122,125) | 46.06 (10.178) | 46.25 (10.955) | 49.10 (9.865)
  Social functioning: Day 85 (n=111,109,121) | 45.89 (11.916) | 46.89 (10.454) | 49.10 (9.581)
  Social functioning: FE (Day155/EW) (n=130,130,127) | 45.81 (11.440) | 46.11 (11.475) | 49.01 (10.521)
  Role-Emotional: Baseline (n=130,130,127) | 51.13 (7.916) | 51.22 (8.515) | 51.20 (8.500)
  Role-Emotional: Day 29 (n=127,122,125) | 48.82 (8.891) | 48.29 (10.837) | 51.69 (8.425)
  Role-Emotional: Day 85 (n=111,109,121) | 49.27 (9.126) | 49.72 (8.104) | 51.60 (7.466)
  Role-Emotional: FE (Day 155/EW) (n=130,130,127) | 48.38 (10.419) | 48.18 (9.941) | 50.80 (8.785)
  Mental health: Baseline (n=130,130,127) | 50.01 (7.632) | 50.34 (8.161) | 50.62 (8.457)
  Mental health: Day 29 (n=127,122,125) | 47.77 (8.793) | 46.33 (10.524) | 52.02 (8.417)
  Mental health: Day 85 (n=111,109,121) | 48.87 (9.402) | 47.18 (9.669) | 51.11 (8.021)
  Mental health: FE (Day 155/EW) (n=130,130,127) | 47.48 (10.270) | 48.19 (9.648) | 51.14 (8.322)

ADVERSE EVENTS:
Arm/Group | Topiramate (JNS019) 50 mg | Topiramate 100 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 2/130 | 4/130 | 2/127
Other Adverse Events (participants affected / at risk) | 125/130 | 121/130 | 106/127
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Topiramate (JNS019) 50 mg (N=130) | Topiramate 100 mg (N=130) | Placebo (N=127)
Shingles (Infections and infestations) | 1 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0
Migraine (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
Closed-angle glaucoma (Eye disorders) | 0 | 1 | 0
Hemorrhagic gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1
Ureterodialysis (Renal and urinary disorders) | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Topiramate (JNS019) 50 mg (N=130) | Topiramate 100 mg (N=130) | Placebo (N=127)
Nasopharyngitis (Infections and infestations) | 45 | 39 | 37
Decreased appetite (Metabolism and nutrition disorders) | 8 | 11 | 3
Paraesthesia (Nervous system disorders) | 38 | 50 | 4
Dysaesthesia (Nervous system disorders) | 35 | 26 | 7
Somnolence (Nervous system disorders) | 21 | 16 | 15
Disturbance in attention (Nervous system disorders) | 7 | 4 | 2
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 13 | 16 | 10
Diarrhoea (Gastrointestinal disorders) | 11 | 7 | 7
Nausea (Gastrointestinal disorders) | 8 | 6 | 5
Malaise (General disorders) | 8 | 8 | 6
Weight decreased (Investigations) | 43 | 51 | 11
Blood bicarbonate decreased (Investigations) | 11 | 15 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The disclosure restriction on PI is that the sponsor can review results communications prior to public release and can embargo communications regarding results for a period as the sponsor requires.